CLINICAL TRIAL: NCT01100619
Title: A Phase 1 Drug-Drug Interaction Study of the Effects of XL184 on the Pharmacokinetics of a Single Oral Dose of Rosiglitazone in Subjects With Solid Tumors
Brief Title: A Drug-Drug Interaction Study of the Effects of XL184 (Cabozantinib) on Rosiglitazone in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL184-008
Record Dates: First submitted 2010-03-22; First posted 2010-04-09 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Papillary Thyroid Cancer; Follicular Thyroid Cancer; Huerthle Cell Thyroid Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Carcinoma, Renal Cell | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects will receive daily XL184, and two single doses of rosiglitazone, 3 weeks apart
  Interventions: Drug: rosiglitazone; Drug: XL184

INTERVENTIONS:
Drug: rosiglitazone — one 4 mg dose as a tablet followed by a second 4 mg dose 3 weeks later
  Other Names: Avandia
Drug: XL184 — dosed with capsules daily

SUMMARY:
The primary objective of this clinical study is to determine whether the inhibition of cytochrome P450 (CYP) isozyme CYP2C8 by XL184 observed in in vitro preclinical studies translates into the potential for clinically significant drug-drug interactions in humans. The study will measure the effect of once daily dosing of XL184 on the pharmacokinetics (PK) of rosiglitazone. The PK of XL184 when combined with rosiglitazone will be evaluated as well.

A specific objective of this study is to determine whether the interaction between XL184 and a drug such as rosiglitazone is sufficiently large enough to necessitate a dosage adjustment when used in combination with XL184, or whether the interaction would require additional therapeutic monitoring.

Rosiglitazone, commonly known as Avandia, is a prescription medicine approved by the FDA used to treat adults with Type 2 (adult-onset or non-insulin dependent) diabetes mellitus (high blood sugar). In this study, subjects will only take 2 doses of rosiglitazone. There is no intention of therapy as a result of taking rosiglitazone in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solid tumor that is metastatic or unresectable and is refractory to or progressed (or relapsed) following standard therapies, or a disease for which no standard therapy exists. Initial enrollment will be limited to differentiated thyroid cancer and renal cell carcinoma. Additional criteria will apply.
* One lesion that is not within a previously radiated field and is measurable on computerized tomography (CT), magnetic resonance imaging (MRI) scan.
* Body mass index (BMI) between 18 and 33 kg/m2.
* Karnofsky Performance Status (≥ 70).
* Adequate organ and marrow function.
* Able to reside in the clinic for two one-day confinement periods in their entirety.
* The subject is willing to refrain from consuming CYP-interacting foods including Seville orange-containing products, grapefruit-containing products, and star fruit-containing products, from 72 hours prior to first dose through the Day 23 Discharge.

Exclusion Criteria:

* Restrictions regarding certain prior treatments will apply.
* The subject has experienced clinically-significant hematemesis or hemoptysis of > 2.5 ml of red blood within 28 days prior to the first dose of study treatment, or other signs indicative of pulmonary hemorrhage within 28 days prior to the first dose of study treatment.
* Not recovered from toxicity due to all prior therapies (ie, return to pre-therapy baseline or Grade ≤ 1).
* Primary brain tumor or brain metastases or spinal cord compression, unless completed radiation therapy ≥ 28 days prior to study. treatment or had surgical resection and is stable without steroid and without anti-convulsant treatment for ≥ 10 days.
* Prothrombin time/International Normalized Ratio (PT/INR) or partial thromboplastin time (PTT) at screening ≥ 1.5 times the laboratory upper limit of normal.
* Uncontrolled, significant intercurrent illness.
* Inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Pregnancy or breastfeeding.
* Human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.
* Allergy or hypersensitivity to components of either of the study treatment (XL184 and rosiglitazone) formulations.
* History of any medical or surgical conditions (eg, stomach or intestinal surgery or resection) that would potentially interfere with or alter the gastrointestinal (GI) absorption, distribution, metabolism, or excretion of the study drug (exceptions: appendectomy, hernia repair, and/or cholecystectomy will be allowed).
* History of, or clinical evidence of, pancreatic injury or pancreatitis, including but not limited to having amylase or lipase levels outside of normal limits.
* Hepatic impaired, ie, with a Child-Pugh score of B or C.
* The subject is being treated with drug(s) that are known to be either extensively metabolized by CYP2C8 (for example rosiglitazone), or inhibitors of either CYP2C8 or CYP3A4, or inducers of CYP3A isozymes.
* The subject has used any prohibited prescription medications or products prior to the first Check-in, or is unable or unwilling to forgo the use of such products from the first Check-in through the Day 23 Discharge, unless deemed acceptable by the investigator.
* Poor peripheral venous access.
* The subject is receiving warfarin (or other coumarin derivatives) at study entry and unable to switch to low molecular weight heparin.
* The subject is receiving dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of XL184 and rosiglitazone | at weekly or twice-weekly visits for the first 4 weeks
  To evaluate the effect of multiple daily doses of XL184 on single dose PK of rosiglitazone

SECONDARY OUTCOMES:
Safety and tolerability of repeated administration of XL184 | at weekly or twice-weekly visits, then every 4 weeks
  To evaluate safety and tolerability of daily oral administration of XL184 and two single doses of rosiglitazone
Pharmacokinetics of XL184 after co-administration of rosiglitazone | at weekly or twice-weekly visits for 4 weeks
  To evaluate the plasma PK of XL184 after a single dose of rosiglitazone

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Choueiri TK, Pal SK, McDermott DF, Morrissey S, Ferguson KC, Holland J, Kaelin WG, Dutcher JP. A phase I study of cabozantinib (XL184) in patients with renal cell cancer. Ann Oncol. 2014 Aug;25(8):1603-8. doi: 10.1093/annonc/mdu184. Epub 2014 May 14. PMID 24827131